CLINICAL TRIAL: NCT03601910
Title: An Open-label, Randomized, Fasted, Single-dose, 2-way Crossover Study to Compare the Pharmacokinetic Characteristics and Safety Between CKD-380 10mg and D308 10mg in Healthy Male Adults
Brief Title: Clinical Study to Compare the Pharmacokinetic Characteristics and Safety Between CKD-380 10mg and D308 10mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 181BE18007
Record Dates: First submitted 2018-07-09; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): 1. Period 1: D308 10mg Tab. 1T
  2. Period 2: CKD-380 10mg Tab. 1T
  Interventions: Drug: D308 10mg Tab.; Drug: CKD-380 10mg Tab.
- B group (Experimental): 1. Period 1: CKD-380 10mg Tab. 1T
  2. Period 2: D308 10mg Tab. 1T
  Interventions: Drug: D308 10mg Tab.; Drug: CKD-380 10mg Tab.

INTERVENTIONS:
Drug: D308 10mg Tab. — D308 10mg Tab.1T single oral administration under fasting condition
Drug: CKD-380 10mg Tab. — CKD-380(Dapagliflozin) 10mg Tab.1T single oral administration under fasting condition

SUMMARY:
This study is an open-label, randomized, fasted, single-dose, 2-way crossover study to compare the pharmacokinetic characteristics and safety between CKD-380 10mg and D308 10mg in healthy male adults.

DETAILED DESCRIPTION:
To healthy male subjects of thirty-four (34), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

Reference drug: D308 10mg Tab. / Test drug: CKD-380 10mg Tab.

Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 45 years old healthy male subject at the screening
2. Subject with a body weight more than 50kg and less than ±20% of ideal body weight at the screening(* Ideal body weight = {Height(cm) - 100}x0.9)
3. Subject who is able to provide written informed consent and decided on his own participation after understanding fully to hear a detailed explanation in the clinical study

Exclusion Criteria:

1. Subject who has a disease or history of clinically significant cardiovascular system, respirator, kidney, endocrine system, blood system, digestive system, central nervous system(CNS), urinary system, musculoskeletal system, psychiatric system or malignant tumor etc.
2. Subject who has a history of gastrointestinal disease or gastrointestinal surgery which can affect investigational product absorption
3. Subject who has hypersensitivity to Investigational product(or additives) or any other medicines or medical history of clinically significant hypersensitivity
4. Subject who is determined unsuitable for clinical studyl participation by Health Examination(Disease, past disease history Physical, vital sign, Electrocardiography, laboratory test etc.) at the screening
5. Subject who has laboratory test results at the screening as below 1) AST or AST > 1.25 times upper limit of normal range 2) Total bilirubin > 1.25 times upper limit of normal range 3) eGFR (estimated Glomerular Filtration Rate) < 60 mL/min/1.73 m2 4) Positive results of HBsAg, Anti-HCV Ab, HIV Ag/Ab and Syphilis reagin test 5) Glucose(under fasting condition) < 50mg/dL or >110mg/dL
6. Subject who has hypersensitivity to investigational product, peanut, or bean
7. Subject with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
8. Subject who shows Systolic Blood Pressure ≥140 or <90 mmHg or Diastolic Blood Pressure ≥90 or <60 mmHg at screening after rest longer than 5 minute at the screening
9. Subject who has history of drug abuse
10. Subject who has too much caffeine and alcohol(Caffeine: > 5 cup/day, Alcohol > 210 g/week) / Smoker(>10 cigarettes/day)
11. Subject who had the Investigational Product(IP) administration at other clinical studies or bioequivalence tests within 90 days prior to the first IP administration
12. Subject who has taken drug-metabolizing enzyme induction and/or inhibition drug(such as barbital, etc.) within 30days prior to the first Investigational Product administration
13. Subject who has donated whole blood within 60 days or component blood within 30days prior to the first Investigational Product administration
14. Subject who has foods containing grapefruit within 7days prior to the first Investigational Product administration
15. Subject who has taken ETC(Ethical The Counter) Drug or herb medicine within 14 days or OTC(Over The Counter) Drug or vitamin supplement within 7 days prior to the first Investigational Product administration
16. Subject who is nat able to have foods containing caffeine, drinking alcohol or Smoking during from 24hours before admission to discharge hospitalization
17. Subject who is not eligible for participation in clinical study by investigator's decision including another reason

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-09-21 (Estimated); Study Completion 2018-11-09 (Estimated)

PRIMARY OUTCOMES:
AUCt of CKD-380 and D308 | Pre-dose(0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
  Area under the CKD-380/D308 concentration in blood-time curve from zero to the final
Cmax of CKD-380 and D308 | Pre-dose(0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 hours
  The maximum CKD-380/D308 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Seunghoon Han, Professor, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul, South Korea